CLINICAL TRIAL: NCT03636750
Title: A Phase 1, Safety, Tolerability and Pharmacokinetic Profile Study of Intravenous Injections of HB002.1T (a Vascular Endothelial Growth Factor Receptor Decoy) in Subjects With Solid Tumor
Brief Title: A Study of Injection HB002.1T in Subjects With Solid Tumor
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Huabo Biopharm Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HB002.1T-01
Record Dates: First submitted 2018-08-06; First posted 2018-08-17 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Solid Tumor

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- HB002.1T 2mg/kg (Experimental): Participants received a 2mg/kg dose of HB002.1T via intravenous injection.
  Interventions: Drug: HB002.1T
- HB002.1T 4mg/kg (Experimental): Participants received a 4mg/kg dose of HB002.1T via intravenous injection.
  Interventions: Drug: HB002.1T
- HB002.1T 8mg/kg (Experimental): Participants received a 8mg/kg dose of HB002.1T via intravenous injection.
  Interventions: Drug: HB002.1T
- HB002.1T 12mg/kg (Experimental): Participants received a 12mg/kg dose of HB002.1T via intravenous injection.
  Interventions: Drug: HB002.1T
- HB002.1T 16mg/kg (Experimental): Participants received a 16mg/kg dose of HB002.1T via intravenous injection.
  Interventions: Drug: HB002.1T
- HB002.1T 20mg/kg (Experimental): Participants received a 20mg/kg dose of HB002.1T via intravenous injection.
  Interventions: Drug: HB002.1T

INTERVENTIONS:
Drug: HB002.1T — HB002.1T is a Vascular Endothelial Growth Factor Receptor Decoy

SUMMARY:
The objectives of this study are to evaluate the safety, tolerability, and pharmacokinetic profile of HB002.1T, a human immunoglobulin Fc fusion protein containing domain 2 and flanking sequence of vascular endothelial growth factor (VEGF) receptor-1 in subjects with solid tumor.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 75 years old of either gender;
* Standard treatment failure, or no standard treatment, or subjects with advanced malignant solid tumors diagnosed by histology or cytology that are not suitable for standard treatment at this stage; there is no limit to the number of treatment options before enrollment;
* Anti-tumor therapy such as radiotherapy, chemotherapy, targeted therapy, endocrine therapy or immunotherapy was not received within 4 weeks before the first treatment of HB002.1T. Mitomycin and nitrosourea were administered for 6 weeks, fluorouracil Oral medications such as tega, capecitabine for at least 2 weeks from the last dose;
* At least one evaluable lesion according to RECIST 1.1;
* ECOG(Eastern Cooperative Oncology Group) performance status 0 or 1
* The expected survival period is not less than 12 weeks;
* The organ function indicated by the following laboratory indicators must be met:

  1. No growth factor support therapy within 14 days, absolute neutrophil count ≥1.5E+9/L;
  2. No transfusion support therapy or growth factor therapy within 14 days , hemoglobin ≥ 90g/L;
  3. Platelet count ≥ 100E+9/L;
  4. Serum creatinine ≤ 1.5 × upper limit of normal (ULN), or creatinine clearance ≥ 60mL / min (serum creatinine > 1.5 × ULN);
  5. Total bilirubin ≤ 1.5 × ULN;
  6. Serum aspartate aminotransferase (AST) and alanine aminotransferase (ALT) concentrations ≤ 2.5 × ULN, or when elevated due to tumor liver metastasis, ALT and AST ≤ 5 × ULN as judged by the investigator;
  7. Electrolyte: blood potassium ≥ 3.0 mmol/L; blood calcium ≥ 2.0 mmol/L;
  8. Prothrombin time (PT) ≤ 1.2 × ULN;
  9. Partial promotion prothrombin time (APTT) ≤ 1.2 × ULN;
  10. Urine test paper test results show that urine protein < 1 +, if ≥ 1 +, need to meet the 24-hour urine protein content <1g.
* The toxicity of previous treatment has been restored to NCI CTCAE ≤ 1 (except for hair loss);
* Women and men of childbearing age must agree to take effective contraceptive measures after signing informed consent, during the study period and within 3 months after the last dose of HB002.1T, and the results of the pregnancy test for women of childbearing age must be negative;
* Subjects must voluntarily sign written informed consent;
* Subjects are able to communicate well with the investigator and are able to comply with research regulations.

Exclusion Criteria:

* Patients with confirmed active central nervous system metastasis and/or cancerous meningitis; but patients with central nervous system metastases who have received treatment and achieved clinical stability for 3 months before starting the study can be enrolled;
* A history of infection with human immunodeficiency virus, or other acquired, congenital disease, or history of organ transplantation;
* Active hepatitis B patients (viral titer is above the upper limit of detection); or hepatitis C virus infection;
* Subjects who have previously been allergic to macromolecular protein preparations/monoclonal antibodies, or known to be allergic to any of the test drug components or excipients;
* Those who have received other clinical trial drugs within 4 weeks before the first treatment of HB002.1T;
* Those who have undergone major surgery within 4 weeks prior to screening;
* Minor surgical procedures (including catheterization, no peripheral venous puncture central catheterization) within 2 days prior to screening; venous puncture center catheterization);
* Patients with systolic blood pressure ≥140mmHg and/or diastolic blood pressure or diastolic blood pressure ≥90mmHg after antihypertensive treatment (one antihypertensive drug is allowed in the baseline period, and the compound preparation is recognized as two);
* The subject has an active infection or during the screening period, the unexplained fever occurs before the first dose > 38.5 °C;
* Those who have had hemoptysis within 4 weeks before screening (defined as coughing with ≥1 teaspoon of blood), but do not rule out cough only with sputum or small blood clot;
* Subjects suffering from the following serious complications:

  1. Unstable angina and/or congestive heart failure or vascular disease requiring hospitalization within 12 months (eg, aortic aneurysm peripheral thrombectomy), or vascular disease (eg, aorta requiring surgical repair) Peripheral static thrombus), other heart damage that the investigator judges is not suitable for clinical trials (eg, poorly controlled arrhythmias, muscle infarction, etc.);
  2. Prior arterial thromboembolic events, venous thrombosis above the venous thrombosis of grade 3 or higher in NCI CTCAE, transient ischemic attack (TIA), cerebral vascular accident (CVA), transmural Myocardial infarction), transmural myocardial infarction, myocardial infarction (MI), hypertensive crisis or encephalopathy; hypertensive crisis or encephalopathy; ), hypertensive crisis or encephalopathy;
  3. Previous or current persistent fulminant hemorrhagic disease;
  4. Chronic Obstructive Pulmonary Disease (COPD) or other respiratory illness requiring hospitalization within 4 weeks prior to screening;
  5. History of abdominal hernia, gastrointestinal perforation abscess or acute bleeding in the first 6 months prior to screening;
  6. Esophageal varices, unhealed wounds or fractures within 6 months prior to screening;
  7. Dominant jaundice and/or caused by abnormal liver function
* Subjects who are in use of warfarin, heparin aspirin (>325 mg/day) or other drugs known to inhibit platelet function within 10 days prior to the first study treatment;
* Subjects receiving dipyridamole, ticlopidine, clopidogrel or cilostazol treatment;
* Subjects with a clear history of neurological or dysfunction, such as poor adherence to epilepsy;
* Pregnant or nursing women;
* Any other reasons assessed by the investigator that are not suitable for participation in the trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2018-06-28 (Actual); Primary Completion 2020-02-20 (Actual); Study Completion 2020-03-21 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) defined as grade 3 or higher National Cancer Institute - Common Terminology Criteria (NCI-CTC) toxicities | 21 days after the first treatment
  Dose-limiting toxicity (DLT) defined as grade 3 or higher National Cancer Institute - Common Terminology Criteria (NCI-CTC) toxicities

SECONDARY OUTCOMES:
Titer and detection rate of anti drug antibody | 1,8,15,and 21 days after the first treatment, at the end of each treatment cycle (cycle 1 is 21 days, cycle 2 to 5 is 14 days) , and and up to 28 days after last treatment
  Titer and detection rate of anti drug antibody
Objective Response Rate | 7 days before first treatment, at the end of treatment cycle 4 and cycle 5 (cycle 1 is 21 days, cycle 2 to 5 is 14 days)
  Objective response rate
Disease Control Rate | 7 days before first treatment, at the end of treatment cycle 4 and cycle 5 (cycle 1 is 21 days, cycle 2 to 5 is 14 days)
  Disease control rate
Computed Tomography | 7 days before first treatment, at the end of treatment cycle 4 and cycle 5 (cycle 1 is 21 days, cycle 2 to 5 is 14 days)
  Computed tomography examination
Peak Plasma Concentration | 1,8,15,and 21 days after the first treatment, at the end of each treatment cycle (cycle 1 is 21 days, cycle 2 to 5 is 14 days) , and and up to 28 days after last treatment
  Peak plasma concentration of patients
Area Under the Plasma Concentration Versus Time Curve (AUC) | 1,8,15,and 21 days after the first treatment, at the end of each treatment cycle (cycle 1 is 21 days, cycle 2 to 5 is 14 days) , and and up to 28 days after last treatment
  Area under the plasma concentration versus time curve (AUC) of patients

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai East Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No